CLINICAL TRIAL: NCT02918942
Title: Tympanoseal (Tympanic Membrane Device) Clinical Study
Status: Completed | Type: Interventional
Sponsor: Grace Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015.01
Record Dates: First submitted 2016-09-26; First posted 2016-09-29 (Estimated); Results first posted 2024-10-15 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-09

CONDITIONS: Tympanic Membrane Perforation
MeSH Terms: conditions — Tympanic Membrane Perforation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | Unapproved Device: Yes

ARMS (1):
- Tympanoseal (Experimental): All subjects will receive the Tympanoseal device.
  Interventions: Device: Tympanoseal

INTERVENTIONS:
Device: Tympanoseal — All subjects will receive the Tympanoseal device that will be placed during a surgical procedure.

SUMMARY:
The purpose of this investigational study is to assess the ability of Tympanoseal (sodium/calcium alginate), an investigational device, to act as a scaffold during healing of the tympanic membrane. Tympanoseal is intended for use following removal or extrusion of indwelling tympanostomy tubes or traumatic injury of the tympanic membrane.

DETAILED DESCRIPTION:
This study will provide data on the safety and the ability of sodium/calcium alginate gels to act as a scaffold capable of occluding a tympanic membrane perforation over the duration of complete healing. Tympanoseal could be used in cases where cartilage or fat graft tympanoplasty would be indicated.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients over 2 years of age at enrollment
* Documentation of a retained tympanostomy tube or persistent perforation less that 5 mm.
* Written informed consent (and assent when applicable) obtained from subject or subject's legal guardian and ability for subject to comply with the requirements of the study

Exclusion Criteria:

* Active otorrhea or otitis media
* History of cholesteatoma
* Perforations on the edge of the tympanic membrane
* Presence of a condition or abnormality that in the opinion of the Investigator would compromise the safety of the patient or the quality of the data
* Subject is taking systemic corticosteroids
* Subject requires continued use of any type of topical otic medication

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2016-10-04 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Plano, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Tympanoseal: All subjects will receive the Tympanoseal device.
  Tympanoseal: All subjects received the Tympanoseal device. Tympanoseal was placed during a surgical procedure.
Period: Overall Study
Arm/Group | Tympanoseal
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tympanoseal
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 25
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 21
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 20
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Serious Adverse Events
Description: The purpose of this investigational study is to assess the safety of Tympanoseal when used during the healing process.
  Subject will be observed during the study and the healing process of the tympanic membrane. Information will be gathered via report forms during regular visits of the patient to the investigator. Any serious adverse events (SAE) will be noted.
  An SAE is defined as any adverse event occurring that results in any of the following outcomes:
  1. Death
  2. A life-threatening adverse experience
  3. An inpatient hospitalization or prolongation of existing hospitalization
  4. A persistent or significant disability/incapacity
  5. A congenital anomaly/birth defect
  6. Required Intervention to Prevent Permanent Impairment or Damage
Time Frame: 16 weeks
Measure: Number; unit: Serious Adverse Event
Arm/Group | Tympanoseal
Number analyzed (Participants) | 25
Serious Adverse Event | 0

2. Secondary Outcome: Number of Participants With Treatment-related Adverse Events
Description: Determine if any adverse events occur during presence of material on tympanic membrane.
Time Frame: 16 weeks
Measure: Number; unit: Participants
Arm/Group | Tympanoseal
Number analyzed (Participants) | 25
Participants | 14

ADVERSE EVENTS:
Time Frame: Adverse event data was gathered at follow up visits which occurred at 4 weeks, 10 weeks, 16 weeks, 20 weeks, 24 weeks, 30 weeks, 36 weeks, 42 weeks, 48 weeks, 54 weeks as needed until the patient exited the study. Follow up visits occurred through study completion, an average of 30 weeks.
Arm/Group | Tympanoseal
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 14/25
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tympanoseal (N=25)
Otorrhea (Ear and labyrinth disorders) | 13 (25)
Granulation (Ear and labyrinth disorders) | 2 (2)
Drainage (Ear and labyrinth disorders) | 3 (3)
Otitis Externa (Ear and labyrinth disorders) | 5 (5)
Otitis Media (Ear and labyrinth disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2017-07-12): https://cdn.clinicaltrials.gov/large-docs/42/NCT02918942/Prot_000.pdf